CLINICAL TRIAL: NCT05681104
Title: Bio-electrical Impedance Analysis and Waist-height Ratio Versus Body Mass Index in Early Detection of Metabolic Syndrome and Obesity Comorbidities in Primary School Aged Obese Children
Brief Title: Early Detection of Metabolic Syndrome and Obesity Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Shawky Ibrahim Abd Elalem, doctor, Assiut University
Other Study IDs: metabolic syndrome in children
Record Dates: First submitted 2022-12-29; First posted 2023-01-12 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Metabolic Disorders in Children
MeSH Terms: interventions — Waist-Height Ratio; Body Mass Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Waist-height ratio — Waist-height ratio as early predictors of metabolic syndrome in primary school obese children
Diagnostic Test: body mass index — Body mass index as early predictors of metabolic syndrome in primary school obese children
Diagnostic Test: Bio-electrical impedance analysis — Bio-electrical impedance analysis as early predictors of metabolic syndrome in primary school obese children

SUMMARY:
To assess :

Compare predictive value of waist to-height ratio and bio-electrical impedance analysis versus BMI in early detection of metabolic syndrome parameters and complication of obesity.

DETAILED DESCRIPTION:
Childhood Obesity is defined as a body mass index (BMI) above the 95th percentile for sex and age.It is Labelled as a national epidemic and affects one in three adults and one in six children in the United States of America.Worldwide several countries have witnessed a double or triple escalation in the prevalence of obesity in the last three decades probably due to urbanization, sedentary lifestyle, and increase consumption of high-Calorie processed food.Based upon the World Population Review 2020, Egypt ranked as the highest 19th country in the world and the 7th highest country in the Arab region, with a 32% obesity rate. In Qena government study was conducted on 1000 students were chosen randomly from all grades of primary schools the overall prevalence of obesity and Overweight was 13.9% and 16.2% respectively. Girls were more obese than boys.

The alarming increase in childhood obesity foreshows a tremendous burden of chronic disease prevention in the future public healthcare systems worldwide. Obesity prevention is a critical factor in controlling Obesity-related Non-communicable diseases (OR-NCDs), including insulin resistance/ metabolic syndrome, coronary artery Disease ,cancer and psychological problems.

Metabolic syndrome is a clustering of abdominal obesity-associated factors including elevated waist Circumference(WC), elevated blood pressure (BP), elevated glucose, elevated triglycerides (TGs) or reduced high-Density lipoprotein cholesterol (HDL-C).two key components of metabolic syndrome glucose and triglycerides are overproduced by the fatty liver. So liver is therefore a key determinant of metabolic abnormalities and prevalence of both metabolic syndrome and Non-alcoholic fatty liver (NAFLD) increases with obesity.

There are various diagnostic methods for metabolic syndrome in children and adolescents. Based on the world Health organization(WHO) criteria it diagnosed when three or more of the following features are found: body Mass index (BMI):>95th percentile, hyperinsulinemia or impaired fasting glucose or impaired glucose tolerance, BP>95th percentile, triglycerides (TG)>105/136 mg/dL (1.2/1.5 mmol/L) for children aged<10 and>10 years Respectively ,high density lipoprotein (HDL)-C<35 mg/dL (0.9 mmol/L).

While BMI is a simple measure calculated by dividing the body weight by the squared height, it does not fully Reflect adiposity or body composition. So a better anthropometric measures than BMI to screen for central obesity are needed. . Among the anthropometric measures used to evaluate adiposity, the waist circumference and waist-To-height ratio (WHtR) can be easily measured in clinical settings and can act as an indicator of central obesity and cardio metabolic risk.

In this study we will Compare predictive value of waist to-height ratio and bio-electrical impedance analysis versus BMI in early detection of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Obese children (Body mass index >95th percentile) aged 6-12 years old

Exclusion Criteria:

Patient who aged <6 or>12 years Presence of chronic illness (diabetes, asthma, endocrine disease) Presence of obesity as a part of genetic syndrome Presence of history of long term drug intake (corticosteroids )

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Obese children (Body mass index >95th percentile) aged 6-12 years old
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
screening tool for metabolic syndrome | At recruitment
  Bio-electrical impedance analysis as an early predictors of metabolic syndrome in primary school obese children

SECONDARY OUTCOMES:
metabolic syndrome diagnostic tool | At recruitment
  Body mass index as an early predictors of metabolic syndrome in primary school obese children

OTHER OUTCOMES:
screening tool | At recruitment
  waist-height ratio as an early predictors of metabolic syndrome in primary school obese children

CONTACTS AND LOCATIONS:
Overall Officials: Ghada om El-sedaffy, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rundle AG, Factor-Litvak P, Suglia SF, Susser ES, Kezios KL, Lovasi GS, Cirillo PM, Cohn BA, Link BG. Tracking of Obesity in Childhood into Adulthood: Effects on Body Mass Index and Fat Mass Index at Age 50. Child Obes. 2020 Apr;16(3):226-233. doi: 10.1089/chi.2019.0185. PMID 32191541
- [Background] Balasundaram P, Daley SF. Public Health Considerations Regarding Obesity. 2025 Feb 15. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK572122/ PMID 34283488
- [Background] Henry FJ. Obesity prevention: the key to non-communicable disease control. West Indian Med J. 2011 Jul;60(4):446-51. PMID 22097676
- [Background] Liang X, Zhang P, Luo S, Zhang G, Tang X, Liu L. The association of quality of life and personality characteristics with adolescent metabolic syndrome: a cohort study. Health Qual Life Outcomes. 2021 Jun 8;19(1):160. doi: 10.1186/s12955-021-01797-7. PMID 34103067